CLINICAL TRIAL: NCT03926702
Title: Tau Imaging With JNJ067
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 073H040
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Progressive Supranuclear Palsy
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Supranuclear Palsy, Progressive | interventions — Radiopharmaceuticals

STUDY DESIGN:
Intervention Model Description: All participants will undergo the same evaluation, which includes screening, cognitive assessment, magnetic resonance imaging scanning (MRI) of the brain, and genetic testing for Apolipoprotein E. Subsequently all subjects will undergo positron-emission tomography (PET) scanning with C-11 PIB (Pittsburgh compound B) for amyloid detection, and JNJ067 for tau detection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiopharmaceutical administration (Experimental): All participants receive radiopharmaceutical for positron-emission tomography (PET) study.
  Interventions: Drug: Radiopharmaceuticals

INTERVENTIONS:
Drug: Radiopharmaceuticals — All subjects will receive radiopharmaceutical for positron-emission tomography (PET) scan.

SUMMARY:
This protocol is designed to assess the utility of a new positron emission tomography (PET) radiopharmaceutical to image tau, [18F] JNJ067, invented by Janssen Pharmaceutical companies of Johnson & Johnson. To date, the radiopharmaceutical has been used in a small group of patients and controls (<20). The study plans to expand the range and number of subjects, to examine a total of 18 participants including controls and patients with Alzheimer's disease (AD) and other dementias. All patients will be recruited from the University of California, San Francisco (UCSF) Memory and Aging Center (MAC) and controls will be recruited from the University of California, Berkeley Aging Cohort Study (BACS). Patients will undergo a multidisciplinary clinical evaluation for diagnosis and a cognitive assessment at the MAC; controls will undergo the usual BACS cognitive assessment performed on the Berkeley campus. Following these evaluations UCSF subjects will undergo magnetic resonance imaging (MRI) scanning at the UCSF Neuroimaging Center and blood sampling for genetic testing also at UCSF, and BACS subjects will undergo an MRI at the University of California Berkeley 3T Brain Imaging Center (in Li Ka Shing hall on the Berkeley campus) and blood sampling for genetic testing at the time of the PET scan.

All subjects will come to Lawrence Berkeley National Law (LBNL) where they will have, on the same day, a C-11 Pittsburgh compound B (PIB) PET scan to measure brain amyloid, and an F-18 JNJ067 PET scan to measure brain tau. These scans will be examined and analyzed by LBNL staff, and data will be processed to examine basic questions about the quantitative behavior of JNJ067. Scan results will not be returned to control subjects, but physicians at UCSF will receive scan results on MAC patients and will share results with participants.

As part of this protocol, the investigators also plan to share the acquired data widely. All data will be de-identified. Data will be shared with the inventors (Janssen/Johnson & Johnson) as well as other scientists worldwide. As this is a new radio tracer, the investigators anticipate that there will be interest in seeing the actual data to answer questions about uptake and application of the method in future studies in many different laboratories. Shared data will include PET scans, MRI scans, genetic testing, and neuropsychological results.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers: Subjects must be aged 50 and over. These individuals will all be of good general medical health with no neurological diseases and capable of providing informed consent.
* Patients: Subjects must be aged 50 and over. Patients will meet diagnostic criteria at UCSF for Alzheimer's disease (AD), mild cognitive impairment (MCI), or progressive supranuclear palsy (PSP).

Exclusion Criteria:

* Any medical contraindications to an MRI scan
* A pacemaker
* Metal clips in brain or tattoos above neck
* Metallic implants or shrapnel in body
* Any body jewelry or piercings that are not removable
* A history of claustrophobia
* A known major systemic disease
* A history of a psychiatric disorder
* A history of substance abuse (prescription or non-prescription) within the past 5 years
* A current weight of less than 45 kilograms (100 pounds)
* Difficulty in urinating or emptying the bladder
* Under age 50
* Participating in an experimental radiotracer study
* Subjects must be fluent English speakers

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Positron-emission tomography (PET) scan results | 3 hours
  PET standard uptake value ratio (SUVR) data

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Possibility to share PET data